CLINICAL TRIAL: NCT04947059
Title: A Prospective Phase III Randomized Clinical Trial Comparing the Effectiveness of Immediate Postoperative Intravesical Instillation With Either Gemcitabine Hydrochloride or Epirubicin Hydrochloride in Patients With Urinary Bladder Cancer (Gemcitabine Epirubicin Normal SAline)
Brief Title: Effectiveness of an Immediate Postoperative Intravesical Instillation With Either Gemcitabine or Epirubicin in Patients With Urinary Bladder Cancer (Gemcitabine Epirubicin Normal SAline)
Acronym: GENSA
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: University of Thessaly (Other)
Responsible Party: Principal Investigator, Vasileios Tzortzis, Professor of Urology, University of Thessaly
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 11006/28.04.2021
Record Dates: First submitted 2021-06-17; First posted 2021-07-01 (Actual); Last update posted 2022-01-26 (Actual); Status verified 2022-01

CONDITIONS: Bladder Cancer
Keywords: Postoperative intravesical instillation; Gemcitabine; Epirubicin
MeSH Terms: conditions — Urinary Bladder Neoplasms

STUDY DESIGN:
Intervention Model Description: Bladder cancer patients, who are treated with a transurethral resection of the bladder tumor, receive postoperatively an immediate single intravesical instillation with either gemcitabine hydrochloride or epirubicine hydrochloride
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Gemcitabine (Active Comparator): Bladder cancer patients, who are treated with a transurethral resection of a bladder tumor, receive postoperatively, within 6 hours after the resection, an immediate single intravesical instillation with gemcitabine hydrochloride 2gr in 100ml of saline for 45-60 minutes and continuous saline irrigation for 24 hours
  Interventions: Drug: Gemcitabine Hydrochloride combined with continuous saline irrigation
- Epirubicin (Active Comparator): Bladder cancer patients, who are treated with a transurethral resection of a bladder tumor, receive postoperatively, within 6 hours after the resection, an immediate single intravesical instillation with epirubicine hydrochloride 50mg in 50ml of saline for 45-60 minutes and continuous saline irrigation for 24 hours
  Interventions: Drug: Epirubicin Hydrochloride combined with continuous saline irrigation

INTERVENTIONS:
Drug: Gemcitabine Hydrochloride combined with continuous saline irrigation — Immediate single intravesical instillation with gemcitabine combined with continuous saline irrigation in bladder cancer patients who are treated with a transurethral resection of the tumor
  Other Names: GROUP A
  Arms: Gemcitabine
Drug: Epirubicin Hydrochloride combined with continuous saline irrigation — Immediate single intravesical instillation with epirubicin combined with continuous saline irrigation in bladder cancer patients who are treated with a transurethral resection of the tumor
  Other Names: GROUP B
  Arms: Epirubicin

SUMMARY:
The natural history of non-muscle-invasive bladder cancer is characterised by recurrence and progression. We compare the effectiveness of gemcitabine hydrochloride and epirubicin hydrochloride, in combination with continuous saline irrigation, as an immediate single intravesical instillation in the potential reduction of the disease recurrence as well as progression.

DETAILED DESCRIPTION:
Bladder cancer (BLCa) is the seventh most commonly diagnosed cancer in the male population worldwide, while it drops to tenth when both genders are considered. At diagnosis about 75% of the patients suffer from non-muscle-invasive BLCa. The natural history of this disease is characterised by recurrence and progression. In order to reduce the possibilities for recurrence, and therefore progression, an immediate single intravesical instillation (ISIVI) of a chemotherapeutic agent has been shown to act by destroying circulating tumour cells after transurethral resection of urinary bladder tumors (TURB), and by an ablative effect on residual tumour cells at the resection site and on small overlooked tumours. Several agents, among them gemcitabine and epirubicin, have been used for the ISIVI so far. Moreover, four large meta-analyses comprising 1,476 to 3,103 patients have consistently shown that after TURB, ISIVI significantly reduces the recurrence rate compared to TURB alone. Furthermore, two meta-analyses suggest efficacy of continuous saline irrigation (CSI) in the prevention of early recurrences. The prevention of tumour cell implantation should be initiated within the first few hours after TURB. After that, tumour cells are firmly implanted and are covered by the extracellular matrix. In all ISIVI studies, the instillation was administered within 24 hours. Until today, no randomised comparisons of individual drugs, combined or not with CSI, have been conducted.

After the initial TURB, the patients will be treated with CSI for 24 hours. Then, they will be randomised, either to gemcitabine or epirubicin, and within 6 hours after the TURB they will receive an ISIVI with gemcitabine or epirubicin, as follows:

- GROUP A: Gemcitabine hydrochloride 2gr in 100ml 0.9% NaCl for 45-60 minutes

- GROUP B: Epirubicin hydrochloride 50mg in 50ml 0.9% NaCl for 45-60 minutes

During the ISIVI the CSI will be stopped.

The ISIVI will not be applied in the following cases:

* Active bleeding, which does not allow to interrupt the CSI
* Postoperative fever > 38°C
* Deep resection of the tumor, which could be associated with bladder perforation and therefore potential extravasation of the administered drug
* Known allergy to gemcitabine or epirubicin

The postoperative follow-up for patients with disease stage pTis, Ta, T1 low grade (LG) / high grade (HG), will be done according to the Guidelines of the European Association of Urology (EAU) for non-muscle-invasive bladder cancer, as follows:

* 1st and 2nd year: Cystoscopy & cytological examination of urine every 3 months, CT Urography every 12 months for HG patients
* 3rd year: Cystoscopy & cytological examination of urine every 6 months, CT Urography every 12 months for HG patients

ELIGIBILITY:
Inclusion Criteria:

* Primary urinary bladder tumor
* Secondary urinary bladder tumor (recurrence)
* Bipolar or monopolar resection
* Creat <2.2mg/dl
* 35% <Hct <52%
* White bloode cells count WBC ≥3000 / μL
* 75000 <PLT <500000 / μL
* Urine culture: negative / sterile
* Alkaline phosphatase, total bilirubin, SGOT, SGPT: values as high as 2 times above the upper normal limit
* Good clinical condition (according to Eastern Cooperative Oncology Group PS ≤ 1)
* CT Urography without findings suggesting an upper urinary tract tumor in the last 3 months before the transurethral resection of the bladder tumor

Exclusion Criteria:

* More than 2 low grade / high differentiation (low grade / LG) histologically confirmed bladder tumors in the last 18 months before the transurethral resection of the bladder tumor
* High grade / low differentiation (HG) histologically confirmed bladder tumor in the last 9 months before the transurethral resection of the bladder tumor
* Those who undergo a transurethral resection of a bladder tumor according to the Guidelines of the European Association of Urology for non-muscle-invasive bladder cancer: incomplete resection of tumor, absence of muscle fibers in the sample with the exception of: Ta / LG-G1, primary Cis and finally, pT1 tumors
* Intravesical instillation of chemotherapeutic agent or BCG in the last 6 months before the transurethral resection of the bladder tumor
* History of non-urothelial bladder cancer
* Stage of disease pT2 (muscle-invasive bladder cancer)
* Presence of a tumor in the urethra
* Upper urinary tract malignancy (present or anamnestically)
* History of pelvic radiotherapy
* Histrory of another malignancy in the last 5 years before the transurethral resection of the bladder tumor

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2021-12-14 (Actual); Primary Completion 2025-10 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Bladder cancer recurrence | At 3 months after the transurethral resection of a bladder tumor
  Histologically proven bladder cancer recurrence
Bladder cancer progression | At 3 months after the transurethral resection of a bladder tumor
  Histologically proven bladder cancer progression
Bladder cancer recurrence | At 12 months after the transurethral resection of a bladder tumor
  Histologically proven bladder cancer recurrence
Bladder cancer progression | At 12 months after the transurethral resection of a bladder tumor
  Histologically proven bladder cancer progression

SECONDARY OUTCOMES:
Bladder cancer recurrence | At 24 months after the transurethral resection of a bladder tumor
  Histologically proven bladder cancer recurrence
Bladder cancer progression | At 24 months after the transurethral resection of a bladder tumor
  Histologically proven bladder cancer progression

CONTACTS AND LOCATIONS:
Overall Officials: Vasileios Tzortzis, Professor, Principal Investigator — Urology Department, University of Thessaly, University Hospital of Larissa, Greece
Locations (1):
- Urology Department, University of Thessaly, University Hospital of Larissa, Larissa, Larissa/Thessaly, Greece

IPD SHARING:
Plan to Share IPD: Yes
All IPD that underlie results in a publication
Supporting Information: Study Protocol
Time Frame: After a publication and for a period of 2 years